CLINICAL TRIAL: NCT03133780
Title: A Comparison of the Sedative Effect of Ketamine and Midazolam During Spinal Anaesthesia for Elective Unilateral Inguinal Hernia Repair: A Randomized Comparative Trial
Brief Title: Sedation During Spinal Anesthesia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Seham Mohamed Moeen Ibrahim, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 42017
Record Dates: First submitted 2017-04-26; First posted 2017-04-28 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Sedation During Spinal Anesthesia
MeSH Terms: interventions — Ketamine; Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketamine (Active Comparator): Patients will receive IV ketamine 0.5 mg/kg diluted in normal saline to a volume of 50 ml over 10 min
  Interventions: Drug: Ketamine
- Midazolam (Active Comparator): Patients will receive IV midazolam 0.03 mg/kg diluted in normal saline to a volume of 50 ml over 10 min
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Ketamine — Patient will receive IV ketamine 0.5 mg/kg diluted in normal saline to a volume of 50 ml over 10 min
  Other Names: Ketalar
  Arms: Ketamine
Drug: Midazolam — Patient will receive IV midazolam 0.03 mg/kg diluted in normal saline to a volume of 50 ml over 10 min
  Other Names: dormicum
  Arms: Midazolam

SUMMARY:
Patients during spinal anesthesia should be sedated.

DETAILED DESCRIPTION:
Spinal anesthesia offers a number of advantages to both the patient and the physician. However, patients are often reluctant to remain awake during a procedure. Sedation has been shown to increase patient satisfaction during regional anesthesia and may be considered as a means to increase the patient's acceptance.Therefore, provision of adequate sedation is important if the advantages of spinal anesthesia are to be fully appreciated.

ELIGIBILITY:
Inclusion Criteria:

* Male patients aged from 18 to 50 years old undergoing elective unilateral inguinal hernia repair with no neurological, cardiovascular and hepato-renal abnormalities.

Exclusion Criteria:

* Age: younger than 18 or older than 50.
* Psychatric or neurological disorders.
* Cardiovascular disorders.
* Coagulation disorders.
* Contraindications to neuraxial block (allergy to L.A, peripheral neuropathy, prior spine surgery).

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2018-07-14 (Actual); Primary Completion 2020-03-07 (Actual); Study Completion 2020-03-07 (Actual)

PRIMARY OUTCOMES:
Time for the onset of sedation in minutes assessed by modified observer's assessment of alertness/sedation score | 90 minutes after spinal anesthesia
  assessed by modified observer's assessment of alertness/sedation score

CONTACTS AND LOCATIONS:
Overall Officials: Seham M Moeen, MD, Principal Investigator — Assiut Univerisity
Locations (1):
- Faculty of Medicine Assuit University, Asyut, Asyut Governorate, Egypt